CLINICAL TRIAL: NCT03813316
Title: Approaches To Therapy Escalation In T2D: A Cluster Randomized Control Trial (ATTACC)
Brief Title: Approaches To Therapy Escalation In T2D
Acronym: ATTACC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding availability to complete project
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Syreon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58214
Record Dates: First submitted 2018-12-24; First posted 2019-01-23 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Type2 Diabetes
Keywords: Diabetes; Type 2; T2D
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate; Sodium-Glucose Transporter 2 Inhibitors; ertugliflozin

STUDY DESIGN:
Intervention Model Description: Model Description" by adding another sentence as follows: "Randomization with be cluster-based by investigator to either standard care or specific individualized training for adding DPP-4 inhibitors and/or SGLT2 inhibitors to metformin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): Adding a DPP-4i (sitagliptin) and/or an SGLT2i (ertugliflozin) to metformin after receiving extra training on individualized care.
  Interventions: Drug: DPP-4 inhibitor; Drug: SGLT2 inhibitor; Drug: SGLT2 inhibitor and DPP-4 inhibitor
- Control Arm (Experimental): Adding a DPP-4i (sitagliptin) and/or an SGLT2i (ertugliflozin) to metformin as per standard care/Diabetes Canada guidelines.
  Interventions: Drug: DPP-4 inhibitor; Drug: SGLT2 inhibitor; Drug: SGLT2 inhibitor and DPP-4 inhibitor

INTERVENTIONS:
Drug: DPP-4 inhibitor — Adding sitagliptin (DPP-4i) add-on using a fixed-dose combination with metformin (Janumet® 50/1000 mg BID).
  Other Names: Sitagliptin
Drug: SGLT2 inhibitor — Adding ertugliflozin (SGLT2i) add-on using a fixed-dose combination with metformin(Segluromet® 2.5/1000 mg BID)
  Other Names: Ertugliflozin
Drug: SGLT2 inhibitor and DPP-4 inhibitor — Adding both a DPP-4i as Fixed dose combination (Janumet) plus SGLT2i ertugliflozin (steglatro) as add-on to metformin.
  Other Names: Ertugliflozin and Sitagliptin

SUMMARY:
Type 2 diabetes mellitus (T2D) is a serious public health challenge which affects more than 9% of Canadians older than 20 years, an estimated prevalence that is anticipated to increase by over 40% in the next decade. The microvascular and macrovascular complications of T2D markedly increase the risks of hospitalization, heart disease, amputation, blindness, end stage renal disease and death, with profound socio-economic consequences for patients, families and society.

Optimal glycemic control is fundamental to the management of T2D, as glycated hemoglobin (A1C) levels > 7.0% are associated with a significantly increased risk of both microvascular and cardiovascular complications. But despite detailed clinical practice guidelines for management of hyperglycemia, glycemic control remains sub-optimal in a large proportion of patients. For example, in over 5000 Canadian diabetic patients managed by primary care physicians (PCPs), more than 50% had an A1C > 7% and more than 20% an A1C > 8%.

For patients not achieving glycemic target on metformin monotherapy and without clinical CVD, Diabetes Canada 2018 Guidelines suggest that the preferred oral antihyperglycemic agents as add-on therapy be either DPP-4 inhibitors or SGLT2 inhibitors if avoidance of hypoglycemia and/or weight gain is a priority. Since most patients with type 2 diabetes would benefit from avoidance of hypoglycemia and/or weight gain, there is clinical rationale for adding DPP-4 inhibitors or SGLT2 inhibitors as oral therapy before considering other oral agents like sulfonylureas or thiazolidinediones. This study is designed to explore the possibility of improving care by providing more precise management guidance to primary care physicians when utilizing DPP-4 inhibitors or SGLT2 inhibitors as add-on therapy to metformin.

DETAILED DESCRIPTION:
This cluster-based study will be conducted in a Primary Care clinical practice setting in Canada. A total of approximately 60 physician practices will be stratified into single (1 PCP) or group (>1 PCP) practices and randomized 1:1 into two arms each consisting of approximately 30 Primary Care practices forming the Interventional arm and the Control arm. The study population will include approximately 600 male and female adult participants living in Canada; who have been diagnosed with T2D; who are being treated for this condition by their PCP; who do not have clinical cardiovascular disease (CVD) and whose eGFR is ≥ 60ml/min; who are receiving metformin at a dose of ≥1500 mg/day as monotherapy for T2D; who are not at the target for glycemic control and whose most recent A1C level is between 7.1 % and 9.0 %. Participant enrollment may be adjusted to ensure balanced distribution of glycemic values at entry across this range between study arms.

All physicians in both arms will receive training on the most current Diabetes Canada 2018 Guidelines for pharmacologic management of type 2 diabetes and the role of DPP-4 inhibitors or SGLT2 inhibitors as add-on therapy to metformin. Physicians in the Interventional arm will receive additional training on specific individualized management for adding DPP-4 inhibitors or SGLT2 inhibitors to metformin. The nature of the additional training will be described separately in a physician training manual. To avoid contamination, only physicians who have been randomized to the Interventional arm will be given access to the physician training manual during the operation of the study, while those physicians randomized into the Control arm will continue to follow their routine clinical practice for utilizing DPP-4 inhibitors or SGLT2 inhibitors as add-on to metformin according to the current Diabetes Canada Practice Guidelines.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years of age or older
4. Previously diagnosed with T2D
5. Have a glycated hemoglobin (A1C) result at Baseline between 7.1% and 9%
6. Have an eGFR value at Baseline ≥60 ml/min/1.73m2
7. Receiving stable (≥ 8 weeks) metformin at a dose of ≥1500 mg/day as monotherapy for T2D
8. Ability to take oral medication and be willing to adhere to the study intervention regimen
9. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration
10. No reason for investigator to suspect they will not tolerate the study medication

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Treated with antihyperglycemic agents other than metformin monotherapy.
2. Known allergies or contraindications to the use of either DPP-4 inhibitors or SGLT2 inhibitors
3. Presence of clinical evidence of cardiovascular disease including a history of heart failure, myocardial infarction, unstable angina, severe atherosclerotic cardiovascular disease on angiography, peripheral arterial disease and/or prior low extremity amputation, revascularization or stroke.
4. Known pregnancy or current lactation
5. Women of child bearing age not willing to use a method of contraception.
6. Febrile illness within 30 days of signing informed consent
7. Treatment with another investigational drug or other intervention within 90 days of signing informed consent
8. Any physical or psychological condition(s) or diagnoses that in the opinion of the treating physician may preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
The percentage of participants achieving an A1C value of ≤ 7% at 24 weeks | 24 Weeks
  This study is designed to test the hypothesis that the provision of physician guidance and specialized training on utilizing DPP-4 inhibitors or SGLT2 inhibitors as add-on to metformin will result in more participants achieving glycemic target at Week 24 when compared to a usual care approach.

SECONDARY OUTCOMES:
The percentage of participants achieving an A1C value ≤ 7% at 12 weeks | 12 weeks
  This secondary endpoint will be the proportion of participants who achieve an A1C value of ≤7%
The absolute reduction in A1C from Baseline at 24 weeks | Week 12 and Week 24.
  This secondary endpoint will be the absolute reduction in A1C values between Baseline and Week 12 / Week 24.
The percentage of participants requiring a change of therapy or rescue therapy at 12 weeks | At 12 weeks
  Change in therapy will be defined as a change from baseline in the medications or doses of these medications used for glycemic control during the 26 weeks of observation for each participant. Rescue therapy will be allowable at any time during the study for urgent clinical need, this should be delayed, if possible, for at least 12 weeks following the administration of the study drugs. At 12 weeks, if A1C is > 9.0%, rescue therapy can be initiated.
Drug tolerability including percentage of participants with hypoglycemic events, and percentage with adverse events.events. | 24 weeks
  Hypoglycemic events will be diagnosed based on symptoms (confirmed by self-monitored blood glucose ≤ 3.9 mmol/L where available) and will be categorized into 4 groups of: (a) severe, ie requiring the assistance of another person, (b) non-severe, ie those that could be self-managed, (c) nocturnal, (d) daytime.
The absolute reduction in FPG from Baseline at 24 weeks | 24 weeks
  This secondary endpoint will be the absolute reduction in FPG values between Baseline and Week 24.
The absolute change in body weight from Baseline at 24 weeks | 24 weeks
  This secondary endpoint will be the absolute change in body weight between Baseline and Week 24.
The absolute change in systolic blood pressure from Baseline at 24 weeks | 24 weeks
  This secondary endpoint will be the absolute change in systolic blood pressure from Baseline to Week 24.
The percentage of participants achieving the composite outcome of A1C ≤ 7.0%, no weight gain and no hypoglycemia at Week 24. | 24 weeks
  This secondary endpoint will be the percentage of participants achieving the composite outcome of A1C ≤ 7.0%, no weight gain and no hypoglycemia at Week 24.
The percentage of participants on statin therapy at 24 weeks | 24 weeks
  This secondary endpoint will be the percentage of participants on statin therapy at Week 24.
The percentage of participants on antihypertensive therapy at Week 24. | 24 weeks
  This secondary endpoint will be the percentage of participants on antihypertensive therapy at Week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Goldenberg, MD, Principal Investigator — LMC Clinical Research Inc.